CLINICAL TRIAL: NCT06152926
Title: Physical Activity and Exercise in Urological Cancers Receiving Immune Check Point Inhibitor Treatment - a Qualitative Study Exploring Patient Perspectives and Experiences
Brief Title: Physical Activity and Exercise in Cancer Immunotherapy Treatment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Nicola Peat, Consultant Physiotherapist, Guy's and St Thomas' NHS Foundation Trust
Other Study IDs: 15438
Record Dates: First submitted 2023-11-22; First posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Physical Activity and Exercise in Cancer Immunotherapy Treatment - Exploratory study of experiences and perceptions — People diagnosed with a urological cancer receiving Immune checkpoint inhibitor treatment at a single centre trust will be invited to either face to face or online video-conference individual interviews (Microsoft teams) according to participant preference.
  Consenting participants will be interviewed via semi-structured interview methods round a topic guide and audio-recorded. Inductive thematic analysis will be conducted to explore participant experiences and perceptions of physical activity and exercise.

SUMMARY:
People who are diagnosed with a cancer commonly experience symptoms that affect day-to-day life, including muscle weakness, pain, tiredness and fatigue. These consequences can make it hard for people to tolerate their medical treatments.

It is well known that regular physical activity or planned exercise can help with these symptoms and significantly improve physical and mental health during cancer treatment. Recent animal studies suggest that exercise training can also reduce the number of cancer cells. For example, exercise training in mice produces more immune cells in the tumour. These immune cells in the tumour contribute to the destruction and reduction of the size of the tumour and are a vital component of effective immunotherapy (cancer treatment that helps your immune system fight cancer). In humans, exercise training and the effect on the immune response in tumours are less understood and is a new area being explored. However, we are aware that most people diagnosed with a cancer are not physically active, and especially not during the treatment period. The aim of this study is to understand the experiences and perceptions of physical activity and exercise in those with cancer receiving immunotherapy treatment (such as immune check point inhibitors (ICI). This will help us to create new practices or change practices to help those with cancer to partake in physical activity and exercise when on treatment.

Participants consenting to take part in the study will be individually interviewed through a semi-structured interview.

DETAILED DESCRIPTION:
Purpose and Design:

Immunotherapy drugs have transformed the landscape of cancer treatment in the last decade. New emerging evidence suggest when integrated with existing cancer treatments, exercise has a positive impact on tumour control, with preclinical studies reporting that exercise suppressed tumour growth and rate of recurrence when delivered as a standalone intervention. However, only 20% of people with cancer do sufficient levels of physical activity (PA) and or exercise to meet national guidelines. These activity levels are anticipated to be even less in those receiving active treatment.

While there is evidence which demonstrates barriers, facilitators and preferences to participation in physical activity and exercise for people with cancer, there is little understanding about these factors in cancer patients receiving active treatments such as immune check point inhibitors (a type of immunotherapy treatment). This is an exploratory study looking into the perspectives and experiences physical activity and exercise in people with cancer receiving immunotherapy treatment. The design implicitly involves people with cancer undergoing immunotherapy treatment.

Recruitment:

Potential participants will be identified by a member of their treating team at clinic outpatient appointments or by the patient self-contacting the research team from flyers and posters seen in outpatient clinics. The study will either be introduced during the same clinic by a member of the patients care team or by the research team via phone, following direct patient enquiry about the study. The purpose of the study will be explained, and the potential participant given an opportunity to ask questions about the proposed study. A patient information sheet will be provided. If interested the potential participant will be provided with a consent form and pre-screening questionnaire.

We project that we will be able to recruit approximately 8-12 participants in 6 weeks (including drop-outs and refusals) for 1:1 interviews. It will take up to 6 weeks to complete all the necessary data collection. Data collection will finish once the projected numbers have been met or data collection saturation achieved.

Consent:

Only participants who can provide fully informed consent will take part in the study. If patients wish to participate, they will be asked to complete the consent form. Patients will have at least 48 hours to consider their participation in the study except for those who request a same day researcher contact and consent process. Contact details for the research team will be provided in the information sheet if the patient wishes to discuss the study further at any time point before or after they complete the consent form. Participants will be told about their right to withdraw from the study at any time without any consequences or disadvantage to them or their medical treatment. It will be emphasised that they are not obliged to give any reason for withdrawal.

Risks, burdens and benefits:

The level of risk is low. Participants may find it distressing to discuss their experience, however, this may be balanced by the psychological benefits of having the discussion. Potential benefits may include time to talk and to focus on the information delivered and what they would like to do with the information.

No direct benefit to participants in the study have been expressed. The study is being carried out to better understand the experiences of physical activity and exercise in people with cancer on immunotherapy treatment, with the hope of improving patients care in the future.

Patient confidentiality and privacy:

The Chief Investigator will preserve the confidentiality of participants taking part in the study and is registered under the Data Protection Act.

Transcripts from the interview will be marked only with a study ID number and audio/digital recordings will be deleted once the analysis has been completed.

All information and data collected will be kept strictly confidential. To ensure privacy and security of personal information, all documentation will use confidential pseudonymised identification numbers for analysis. Identification numbers and details of the participant (e.g.name) will be kept on a password protected document and held separately from data. Patients who participate in an interview will be given a pseudonym and will be referred to by this pseudonym in transcripts, the analysis and final reports e.g. when quoting participants. In accordance with the Data Protection Act (2018), electronic data will be stored on a password protected share drive (GSTT NHS Trust secure server) accessible only to the research team. No identifiable information will be used in the reporting of the data.

If it is necessary to break confidentiality due to the participant being at serious risk (ie risk of self harm or harm to others), the clinical nurse specialist or medical team member involved in their care will be informed. Potential risks:

Participants may become distressed during the interviews due to the subject matter. In the event of this happening, the researchers, (who have experience in dealing with sensitive issues) will use their skills and expertise to support the participant. If necessary the interview will be stopped. If needed, a referral can be made to the relevant nurse specialist team who may refer the patient onto the psychological support services. The participant will be given the researchers contact details to make contact if they have any concerns or questions following the interview.

Conflict of interest:

There are no perceived conflict of interest nor significant barriers to impartiality.

Participants will be asked whether they would like to receive a written summary of the findings of the study (sent by email or post according to their preference). Participants can alternatively choose to be informed of the study findings at a future 'Patient' engagement event.

ELIGIBILITY:
Inclusion Criteria:

* Primary Urological (Bladder and Renal) cancer diagnosis receiving or planned immune check point inhibitor treatment at GSTT hospital.
* Adults aged 18 years or older
* Willing and able to take part in Face to Face interviews at a hospital site or virtual video interviews at home.
* Cancer survival >6 month
* Proficient in English

Exclusion Criteria:

* Aged lower than 18 years
* Inability to give informed consent and information (due to unable to speak or understand English)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with a urological cancer (Bladder or Renal) that are receiving or planned to receive immunotherapy treatment (with immune check point inhibitors) at a single centre.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2023-12-04 (Estimated); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Exploration of experiences | 3-6 months
  To understand participant's perspectives and experiences of physical activity and exercise on immune check point immunotherapy treatment through Inductive thematic analysis of semi-structured individual interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Mieke Van-Helmerijk, Study Chair — King's College London

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be disclosed to any other researchers. Participant data from the study will be anonymised and reported within a report for researchers and the general public to review as a peer review report.

REFERENCES:
- [Result] Handford J, Chen M, Rai R, Moss CL, Enting D, Peat N, Karagiannis SN, Van Hemelrijck M, Russell B. Is There a Role for Exercise When Treating Patients with Cancer with Immune Checkpoint Inhibitors? A Scoping Review. Cancers (Basel). 2022 Oct 14;14(20):5039. doi: 10.3390/cancers14205039. PMID 36291823